CLINICAL TRIAL: NCT06946693
Title: Comparative Assessment of the Color Stability and Surface Roughness of Implant-Supported Provisional Restorations Fabricated by Conventional Technique, Milling and 3D Printing: A Randomized Controlled Clinical Trial.
Brief Title: Surface Topography and Color Stability of Conventional, 3D Printed, and Milled Provisional Restorations.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Comparative assessment of the Color Stability and Surface Roughness of Implant-Supported Provisional Restorations Fabricated by Conventional Technique, Milling and 3D Printing: A Randomized Controlled Clinical Trial, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dr. NANG NALIKA MOUNGKHOM
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant
Keywords: PROVISIONAL RESTORATIONS
MeSH Terms: interventions — Printing, Three-Dimensional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- To evaluate the surface roughness and color stability of Conventional provisional restorations (Active Comparator)
  Interventions: Procedure: To evaluate the color stability and surface roughness of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing in mandibular posterior region.
- To evaluate the surface roughness and color stability of 3D Printed provisional restorations (Active Comparator)
  Interventions: Procedure: To evaluate the color stability and surface roughness of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing in mandibular posterior region.
- To evaluate the surface roughness and color stability of Milled provisional restorations (Active Comparator)
  Interventions: Procedure: To evaluate the color stability and surface roughness of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing in mandibular posterior region.

INTERVENTIONS:
Procedure: To evaluate the color stability and surface roughness of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing in mandibular posterior region. — Subjects with single stage implant placement and early non-functional loading with implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing.

SUMMARY:
Patient attending the Outdoor Patient Department of the Department of Prosthodontics at Post Graduate Institute of Dental Sciences, Rohtak will be screened. The screening will include history, consent taking and clinical examination of the partially edentulous patients. Patients will be selected according to the inclusion and exclusion criteria. Single stage endosseous implants will be placed. Provisional restorations fabricated by conventional technique, milling, and 3D printing will constitute three groups, followed by evaluation of color stability and surface roughness after intraoral use.

DETAILED DESCRIPTION:
Title: "Comparative assessment of the color stability and surface roughness of implant-supported provisional restorations fabricated by conventional technique, milling, and 3D printing: A randomized controlled clinical trial" Rationale: The study needs to verify the color stability and surface roughness of implant-supported provisional restorations fabricated using conventional technique, milling, and 3D printing.

Aim and objectives: To evaluate the color stability and surface roughness of implant-supported provisional prosthesis fabricated using conventional technique, milling, and 3D printing in the mandibular posterior region.

Setting: Department of Prosthodontics and Crown & Bridge, PGIDS, Rohtak. Study Design: Randomized controlled clinical trial. Population/Participants: Provisional restoration will be fabricated using conventional technique, milling and 3D printing.

Sample Size: Total of 36 samples will be prepared (n = 12 samples per test group).

Methodology: This is an in-vivo study and will be carried out in the Department of Prosthodontics and Crown & Bridge, Post Graduate Institute of Dental Sciences, Rohtak with the purpose to evaluate the color stability and surface roughness of implant-supported provisional restorations fabricated using conventional technique, milling, and 3D printing in the mandibular posterior region.

Outcome Measures: Measuring the color stability using spectrophotometer and surface roughness using profilometer.

Statistical Analysis: Data obtained will be compiled on MS Office Excel Sheet (v 2010) and will be subjected to statistical analysis using statistical package for social sciences (SPSS v 21.0, IBM). Intergroup and intragroup comparisons will be done according to the distribution of data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects consented to participate in the study. 2. Subjects with maintainable oral hygiene. 3. Subjects with adequate edentulous space at the prospective implant site. 4. Subjects with availability of adequate quantity and quality of bone.

-

Exclusion Criteria:

1. Subject with presence of infection around proposed site of implant placement.
2. Subjects with any condition that would interfere with the soft tissue and bone healing.
3. Subjects in which surgical procedure is contraindicated for any reason.

   -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-18 (Estimated); Primary Completion 2026-08-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Surface roughness of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing. | 1 year 6 months
  Surface roughness of provisional restorations will be measured using profilometer
Color stability of implant supported provisional restorations fabricated using conventional technique, milling, and 3D printing. | 1 year 6 months
  Color stability of provisional restorations will be measured using spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: NALIKA MOUNGKHOM, BACHELOR OF DENTAL SURGERY, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES ROHTAK, HARYANA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No